CLINICAL TRIAL: NCT04588402
Title: Assessing the Population Level Impact of HPV Vaccination on Prevention of Cervical HPV Infection in Sikkim, India
Brief Title: Impact of HPV Vaccination on Prevention of Cervical HPV Infection in Sikkim, India
Acronym: HPV-Vac-S
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Department of Health and Family welfare, Government of Sikkim (Unknown); Sikkim Manipal Institute (Unknown); Rajiv Gandhi Centre for Biotechnology (Industry)
Responsible Party: Sponsor
Other Study IDs: SMIMS/IEC/C/2020-09
Record Dates: First submitted 2020-09-25; First posted 2020-10-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: The study being observational in nature, there is no intervention. The investigators will only collect cervical samples from married women within a specified age range at different intervals. — Women will be approached one time only, when they will attend the gynecology out-patients department for various reasons. After signing the informed consent, the participants will fill in a risk factor questionnaire to study the socio-demographic information, sexual history and HPV vaccination history and the determinent of HPV infection. The questionnaire will be administered by a trained social worker or nurse.
  A gynecologist will collect cervical cells from the participant's cervix during a gynecological examination. The cervical specimen will be examined for presence of specific HPV genotypes and Chlamydia infection.

SUMMARY:
This project aims is to monitor the effectiveness of HPV vaccination in real-word conditions, at least 7 years after initiation of HPV vaccination in Sikkim. This study would give an opportunity to provide rapid feedback to the Indian public health authorities about the impact of the HPV vaccine.

DETAILED DESCRIPTION:
The investigators would like to estimate the prevalence of HPV infections based on cervical samples collected from the Sikkimese women aged 18 to 22 years at baseline (i.e. when the study participants are expected to have no benefit of vaccination) and seven years after the launch of the HPV vaccination programme, by which time the initial vaccinated cohorts will be aged 18 to 22 years and many of them will be sexually active. If the vaccination programme continues with the current high coverage rate, the cohort of women in the second age group are expected to be protected due to herd immunity, irrespective of whether any individual woman receives the vaccine or not. Overall effectiveness to protect women aged 18-22 years against targeted and non-targeted HPV infections will be monitored through repeated cervical sample -based surveys.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 22 years, resident of Sikkim and married.
* Pregnancy will not be considered as exclusion criteria.
* Sample collection should be avoided during active menstruation.

Exclusion Criteria:

* Women who do not provide written consent
* Women who are not able to cooperate in collection of cervical cell sample or respond to questions due to any acute or severe mental and physical illnesses.
* Women who had undergone hysterectomy.
* Vaccinated in research project

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women will be approached one time only, when they will attend the gynecology out-patients department for various reasons.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The reduction in the point prevalence of genotype-specific HPV infection in women within 7 years of initiation of HPV vaccination compared to that at baseline | 7 years
  The investigators will estimate difference in the prevalence of genotype-specific HPV infection based on cervical samples collected from the married women aged 18 to 22 years at baseline (in the year 2020-21) and again in the year 2025-26 (seven years after the initiation of the HPV vaccination program).
The difference in the point prevalence of chlamydia trachomatis infection in women within 7 years of initiation of HPV vaccination compared to that at baseline | 7 years
  The investigators will estimate difference in the prevalence of chlamydia trachomatis infection based on cervical samples collected from the married women aged 18 to 22 years at baseline (in the year 2020-21) and again in the year 2025-26 (seven years after the initiation of the HPV vaccination program). The estimate will allow the investigators to understand any change in the background risk of sexually transmitted infection in the population over time.

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Verma, MD, Principal Investigator — Sikkim Manipal Inst., Sikkim, India; Phumzay Denzongpa, MD, Principal Investigator — Dept of H & FW, Govt. of Sikkim, India
Locations (1):
- Sikkim Manipal Hospital, Gangtok, Sikkim, India

IPD SHARING:
Plan to Share IPD: No